CLINICAL TRIAL: NCT00341172
Title: Discovery of Genetic Variants Contributing to the Incidence or Course of CMV Disease in AIDS Patients
Brief Title: The Effects of Genetic Differences Among AIDS Patients on Cytomegalovirus Retinitis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905023; 05-C-N023
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: AIDS
Keywords: Retinitis; Cytomegalovirus; HIV-1; Polymorphisms; HAART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Retinitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
This study will evaluate the role of certain gene variants on the onset and course of cytomegalovirus (CMV) retinitis-a severe infection affecting the eye-in patients with AIDS. Symptoms include blurry vision, eye pain, photophobia, floaters, eye redness, and impaired vision. Left untreated, it can cause blindness. The study is done in collaboration with investigators of the Longitudinal Studies of the Ocular Complications of AIDS (LSOCA) at the Johns Hopkins University School of Medicine. The purpose of the LSOCA study is to learn about how HIV and other infections associated with AIDS and their treatments affect people's eyes and sight.

Blood samples previously collected from patients participating in the LSOCA study will be analyzed for gene variants. These differences will then be correlated with the patients' clinical data to try to discover the role of gene differences among patients on the following: susceptibility to CMV and related problems; development and course of CMV; and response to HAART (highly active antiretroviral treatment), particularly in CMV onset and pathology.

The study will use blood samples and clinical information previously collected from patients during their participation in LSOCA. The materials will be identified with a numerical code linking the samples and clinical data. No additional procedures will be performed on patients for this study.

DETAILED DESCRIPTION:
Background:

LSOCA is a prospective observational study of ocular complications in HIV-infected AIDS patients including those treated with highly active anti-retroviral treatment (HAART).

In the absence of HAART, there is a 30% risk of cytomegalovirus (CMV0 infection associated with AIDS.

Of these CMV patients, 75-85% will develop retinitis.

Objectives:

Test a number of human candidate gene polymorphisms in the LSOCA cohort samples to discover genetic influences on the susceptibility to CMV and associated pathologies.

Inspect the role of known AIDS restriction genes (ARGs) on the infection and pathogenesis of CMV.

Evaluate the role of the same host gene polymorphisms on the response to HAART, particularly in CMV onset and pathology.

Eligibility:

Lymphocytes for DNA extraction and relevant clinical data from properly consented AIDS patients (maximum estimated at n= 2,000) will be provided to the LGD for genotyping and analysis. No available subjects will be excluded.

Design:

LSOCA has collected blood specimens and banked viably frozen lymphocytes from each study participant. Samples and clinical data are coded and linked.

Genes under study include the traditional described ARGs (O'Brien & Nelson, 2004); the CMV receptor gene, US28 (Pleskoff et al., 1997); HLA class I and II; KIR gene family and other genes involved in virus immune defenses.

Single nucleotide variants within coding regions, upstream and downstream regulatory regions, and ironic elements will be tested for genetic equilibrium distortion in patient populations at risk for CMV and displaying CMV pathology.

Following this study, the samples will be maintained in our repository and curated through our central Laboratory database. Loss or destruction of these samples will be recorded in our database and cannot impact the study participants in any way. We understand that studies subsequent to the completion of this protocol will require additional OHSR/IRB approval prior to commencement.

ELIGIBILITY:
* INCLUSION CRITERIA:

Lymphocytes for DNA and relevant clinical data from properly consented subjects will be provided to the LGD for genotyping and analysis. No available subjects will be excluded.

Diagnosis of AIDS according to the 1993 CDC diagnostic criteria (with or without clinical symptoms of CMV retinitis or other ocular complications of AIDS).

Age 13 years or older

Signed consent statement

For minors, ages 13-17, signed Consent Statement (by parent/guardian) and Assent Statement (by adolescent and parent/guardian).

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CMV Disease in AIDS cohort@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 2232 (Actual)
Dates: Start 2004-10-26 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Collection of 2500 samples | Annually
  this study is complete

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W McVicar, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] O'Brien SJ, Nelson GW, Winkler CA, Smith MW. Polygenic and multifactorial disease gene association in man: Lessons from AIDS. Annu Rev Genet. 2000;34:563-591. doi: 10.1146/annurev.genet.34.1.563. PMID 11092839
- [Background] O'Brien SJ, Moore JP. The effect of genetic variation in chemokines and their receptors on HIV transmission and progression to AIDS. Immunol Rev. 2000 Oct;177:99-111. doi: 10.1034/j.1600-065x.2000.17710.x. PMID 11138790
- [Background] Jabs DA, Van Natta ML, Kempen JH, Reed Pavan P, Lim JI, Murphy RL, Hubbard LD. Characteristics of patients with cytomegalovirus retinitis in the era of highly active antiretroviral therapy. Am J Ophthalmol. 2002 Jan;133(1):48-61. doi: 10.1016/s0002-9394(01)01322-8. PMID 11755839